CLINICAL TRIAL: NCT00983424
Title: A Phase I, Open-label, Study of the Safety and Tolerability of Cyclosporine A (CsA) in Combination With Nab-paclitaxel in Patients With Metastatic Breast Cancer
Brief Title: Cyclosporine A in Combination With Nab-Paclitaxel in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Avon Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 08B7; STU00015585; NCI-2011-00223 (Other: NCI CTRP#)
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclosporins; Cyclosporine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): Cyclosporine A + nab-paclitaxel
  Interventions: Drug: Cyclosporins; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: Cyclosporins — dose escalation, administered orally twice a day
  Other Names: Neoral; Gengraf
Drug: nab-paclitaxel — 100 mg/m2 IV days 1, 8 and 15

SUMMARY:
The purpose of this research study is to evaluate the safety of therapy with nab-paclitaxel and CsA and if the addition of Cyclosporine A (CsA) to nab-paclitaxel helps stop cancer cells as well as or better than nab-paclitaxel alone.

DETAILED DESCRIPTION:
Treatment for metastatic breast cancer commonly involves the use of the chemotherapy drug nab-paclitaxel. Nab-paclitaxel is a special preparation of paclitaxel inside a protein layer of albumin. Other studies have shown Cyclosporine A (CsA) may block the progression of advanced breast cancer. The combination of nab-paclitaxel and CsA is considered investigational which means it has not been approved by the US Food and Drug Administration, FDA. Participants on this study will receive nab-paclitaxel through a vein in the arm weekly 3 weeks out of 4, in the outpatient clinic. On the same day as the first infusion of nab-paclitaxel, participants will begin taking CsA tablets twice a day by mouth. Participants will continue to receive study treatment as long as their tumor responds. If the tumor does not respond or the participant experience severe side effects from study treatment, she will be removed from the study and offered other therapies, if that is appropriate.

ELIGIBILITY:
Inclusion Criteria

* Female or male patients with adenocarcinoma of the breast with metastatic disease.
* Patients may have evaluable or measurable disease.
* Age > 18 years.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Able to swallow and retain oral medication.

Exclusion Criteria

* Patients who have had any major surgery, hormonal therapy (other than replacement), chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Prior nab-paclitaxel is allowed.
* Patients may not be receiving any other investigational agents or receiving concurrent anticancer therapy.
* Patients with uncontrolled brain metastases or leptomeningeal disease or active neurologic impairment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Cyclosporine A or nab-paclitaxel.
* Pregnant or lactating (Cyclosporine A is excreted into breast milk) females
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
* HIV-positive patients are excluded since Cyclosporine A may result in further immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability and feasibility of the combination of Cyclosporine A and nab-paclitaxel in the treatment of metastatic breast cancer (MBC). | labs drawn weekly
To determine the maximum-tolerated dose (MTD) of Cyclosporine A and nab-paclitaxel in patients. | at study completion (estimated at 2 years)

SECONDARY OUTCOMES:
To describe any preliminary evidence of efficacy of Cyclosporine A and nab-paclitaxel in combination in patients. | every 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Gradishar, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Northwestern Medical Faculty Foundation, Chicago, Illinois, United States